CLINICAL TRIAL: NCT02101853
Title: Risk-Stratified Randomized Phase III Testing of Blinatumomab (NSC#765986) in First Relapse of Childhood B-Lymphoblastic Leukemia (B-ALL)
Brief Title: Blinatumomab in Treating Younger Patients With Relapsed B-cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00631; NCI-2014-00631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s15-00970; COG-AALL1331; AALL1331 (Other: Children's Oncology Group); AALL1331 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2022-12-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Stem Cell Transplantation; Asparaginase; Leyk; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Mitoxantrone; pegaspargase; Radiotherapy; Radiation; Hydrocortisone; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (HR and IR control) (Active Comparator): Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, and then undergo allogeneic HSCT. Closed effective September 18, 2019.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Asparaginase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Mitoxantrone; Drug: Mitoxantrone Hydrochloride; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Therapeutic Hydrocortisone; Drug: Vincristine; Drug: Vincristine Sulfate
- Arm B (HR and IR blinatumomab) (Experimental): Patients receive Blinatumomab Block 1 over 5 weeks, Blinatumomab Block 2 over 5 weeks, and then undergo allogeneic HSCT.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: Blinatumomab; Drug: Cytarabine; Drug: Dexamethasone; Drug: Methotrexate; Other: Pharmacological Study; Drug: Therapeutic Hydrocortisone
- Arm C (LR control) (Active Comparator): Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, Continuation 1 over 8 weeks, Continuation 2 over 8 weeks, and then Maintenance.
  Interventions: Drug: Asparaginase; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Pharmacological Study; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine; Drug: Vincristine Sulfate
- Arm D (LR blinatumomab) (Experimental): Patients receive Block 2 over 4 weeks, Blinatumomab Cycle 1 over 5 weeks, Continuation 1 over 8 weeks, Blinatumomab Cycle 2 over 5 weeks, Continuation 2 over 8 weeks, Blinatumomab Cycle 3 over 5 weeks, and then Maintenance.
  Interventions: Biological: Blinatumomab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Leucovorin Calcium; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Pharmacological Study; Radiation: Radiation Therapy; Drug: Therapeutic Hydrocortisone; Drug: Thioguanine; Drug: Vincristine; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HSCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
  Arms: Arm A (HR and IR control); Arm B (HR and IR blinatumomab)
Drug: Asparaginase — Given IM or IV
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine Amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
  Arms: Arm A (HR and IR control); Arm C (LR control)
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
  Arms: Arm B (HR and IR blinatumomab); Arm D (LR blinatumomab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)
Drug: Cytarabine — Given IT and IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)
Drug: Leucovorin Calcium — Given IV or PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
  Arms: Arm C (LR control); Arm D (LR blinatumomab)
Drug: Methotrexate — Given IT, IV, and PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Mitoxantrone — Given IV
  Other Names: Dihydroxyanthracenedione; Mitozantrone
  Arms: Arm A (HR and IR control)
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
  Arms: Arm A (HR and IR control)
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)
Other: Pharmacological Study — Correlative studies
Radiation: Radiation Therapy — Undergo cranial radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm C (LR control); Arm D (LR blinatumomab)
Drug: Therapeutic Hydrocortisone — Given IT
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; Hydrocortisone; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Arm C (LR control); Arm D (LR blinatumomab)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm A (HR and IR control); Arm C (LR control); Arm D (LR blinatumomab)

SUMMARY:
This randomized phase III trial studies how well blinatumomab works compared with standard combination chemotherapy in treating patients with B-cell acute lymphoblastic leukemia that has returned after a period of improvement (relapsed). Immunotherapy with blinatumomab may allow the body's immune system to attack and destroy some types of leukemia cells. It is not yet known whether blinatumomab is more effective than standard combination chemotherapy in treating relapsed B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare disease free survival (DFS) of high-risk (HR) and intermediate-risk (IR) relapse B-cell acute lymphoblastic leukemia (B-ALL) patients who are randomized following induction block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR randomization) as a part of a treatment regimen prior to allogeneic bone marrow transplantation. (Closed to enrollment effective September 18, 2019) II. To compare the DFS of low risk (LR) relapse B-ALL patients who are randomized following block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR randomization). (Closed to enrollment effective September 30, 2019)

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) of HR and IR relapse B-ALL patients who are randomized following induction block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR randomization). (Closed to enrollment effective September 18, 2019) II. To compare OS of LR relapse B-ALL patients who are randomized following block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR randomization).

EXPLORATORY OBJECTIVES:

I. To compare the rates of minimal residual disease (MRD) >= 0.01% at the end of block 2 and block 3 for HR and IR relapse B-ALL patients in HR/IR randomization.

II. To estimate, for treatment failure (TF) patients not previously receiving blinatumomab, the hematologic complete remission rate (CR), rate of MRD < 0.01%, and proportion able to proceed to hematopoietic stem cell transplant (HSCT) in CR after treatment with blinatumomab.

III. To assess the feasibility and safety of rapid taper of immune suppression for the subset of HSCT patients with MRD >= 0.01% pre- and/or post-HSCT with no acute graft versus host disease (aGVHD).

IV. To evaluate blinatumomab pharmacokinetics (PK) and explore exposure-response relationships for measures of safety and effectiveness.

OUTLINE:

All patients receive Block 1 over 4 weeks.

BLOCK 1: Patients receive dexamethasone orally (PO) twice daily (BID) or intravenously (IV) on days 1-5 and 15-19; vincristine sulfate IV over 1 minute on days 1, 8, 15, and 22; pegaspargase IV over 1-2 hours on days 3 and 17; mitoxantrone hydrochloride IV over 15-30 minutes on days 1-2, and methotrexate intrathecally (IT) on day 1. Patients with central nervous system (CNS) 1 or CNS2 also receive methotrexate IT on day 8. Patients with CNS3 (including isolated CNS relapse) also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on days 8, 15, and 22. High risk and intermediate risk patients are then assigned to randomization R1. Low risk patients are assigned to randomization R2.

RANDOMIZATION R1 (HR and IR patients): Patients are randomized to 1 of 2 treatment arms. Effective 09/18/2019, HR/IR patients not yet randomized are not eligible for post-Induction therapy on AALL1331 and will be removed from protocol therapy. Patients receiving therapy on Arm A prior to Amendment #10A who have not yet received day 22 treatment on Block 3 will be offered the opportunity to cross over to Arm B to receive blinatumomab.

ARM A: Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, and then undergo allogeneic HSCT if eligible. Patients with persistent testicular involvement after Block 1 receive testicular radiation during the Block 2.

ARM B: Patients receive Blinatumomab Block 1 over 5 weeks, Blinatumomab Block 2 over 5 weeks, and then undergo allogeneic HSCT if eligible. Patients with persistent testicular involvement after Block 1 receive testicular radiation during the first block of blinatumomab.

RANDOMIZATION R2 (LR patients): LR patients are randomized to 1 of 2 treatment arms.

ARM C: Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, Continuation 1 over 8 weeks, Continuation 2 over 8 weeks, and then Maintenance. CNS3 patients receive chemoradiation post-Maintenance Cycle 1. Patients with persistent testicular involvement after Block 1 receive testicular radiation during Block 2.

ARM D: Patients receive Block 2 over 4 weeks, Blinatumomab Cycle 1 over 5 weeks, Continuation 1 over 8 weeks, Blinatumomab Cycle 2 over 5 weeks, Continuation 2 over 8 weeks, Blinatumomab Cycle 3 over 5 weeks, and then Maintenance. CNS3 patients receive chemoradiation post Maintenance Cycle 1. Patients with persistent testicular involvement after Block 1 receive testicular radiation during Block 2.

BLOCK 2: Patients receive dexamethasone PO BID or IV on days 1-5; vincristine sulfate IV over 1 minute on day 1; methotrexate IV over 36 hours on day 8; leucovorin calcium IV or PO on days 10-11; pegaspargase IV over 1-2 hours on day 9 or 10; cyclophosphamide IV over 15-30 minutes on days 15-19; and etoposide IV over 1-2 hours on days 15-19. Patients with CNS1 or CNS2 also receive methotrexate IT on day 8. Patients with CNS3 also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on days 8 and 22.

BLOCK 3: Patients receive dexamethasone PO BID or IV on days 1-5; vincristine sulfate IV over 1 minute on day 1; cytarabine IV over 3 hours every 12 hours on days 1, 2, 8, and 9; asparaginase intramuscularly (IM) or IV over 1 hour on days 2, 4, 9, 11, and 23; methotrexate IT on day 1and IV over 36 hours on day 22; leucovorin calcium PO or IV on days 24-25. Patients with CNS1 or CNS2 also receive methotrexate IT on day 22. Patients with CNS3 also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on day 22.

BLINATUMOMAB BLOCK 1: Patients receive dexamethasone PO or IV on day 1 and blinatumomab IV continuously on days 1-28. Patients with CNS1 or CNS2 also receive methotrexate IT on days 15 and 29. Patients with CNS3 also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on days 15 and 29.

BLINATUMOMAB BLOCK 2: Patients receive blinatumomab IV continuously on days 1-28. Patients with CNS1 or CNS2 also receive methotrexate IT on days 8 and 29. Patients with CNS3 also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on days 8 and 29.

BLINATUMOMAB BLOCK 3: Patients receive blinatumomab IV continuously on days 1-28 and dexamethasone PO or IV on day 1.

CONTINUATION 1 & 2: Patients receive dexamethasone PO BID or IV on days 1-5; vincristine sulfate IV over 1 minute on day 1; mercaptopurine tablet PO on days 1-42; methotrexate PO on days 8, 15, 29, and 36; or; cyclophosphamide IV over 15-30 minutes on days 43 and 50; etoposide IV over 1-2 hours on days 43 and 50; thioguanine PO once daily on days 43-49; and cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 44-47 and 51-54. Patients with CNS1 or CNS2 also receive methotrexate IT on days 1 and 43, methotrexate PO every 6 hours for 4 doses on day 22, leucovorin calcium PO every 6 hours for 2 doses on day 24. Patients with CNS3 also receive methotrexate IT, hydrocortisone IT, and cytarabine IT on days 1 and 43 ; methotrexate IV over 36 hours on day 22; and leucovorin calcium IV or PO every 6 hours on days 24-25.

MAINTENANCE: Patients receive dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61; vincristine sulfate IV over 1 minute on days 1, 29, and 57; mercaptopurine tablet PO on days 1-84; and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Patients with CNS1 or CNS2 also receive methotrexate IT on day 1. Patients with CNS3 receive Triple Intrathecal Therapy (ITT) on day 1. Cycles repeat every 12 weeks for up to 2 years from the beginning of treatment in the absence of disease progression or unacceptable toxicity.

MAINTENANCE CHEMORADIATION (LR CNS3 PATIENTS ONLY): Following maintenance cycle 1, patients receive 1800 cGy cranial radiation; dexamethasone PO BID or IV on days 1-7 and 15-21; vincristine sulfate IV over 1 minute on days 1, 8 and 15; and pegaspargase IV over 1-2 hours on day 1. Patients then resume maintenance with cycle 2 and beyond.

After completion of study treatment, patients are followed up annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 1 year and < 31 years of age at the time of relapse will be eligible
* First relapse of B-ALL, allowable sites of disease include isolated bone marrow, combined bone marrow and CNS and/or testicular, and isolated CNS and/or testicular; extramedullary sites are limited to the CNS and testicles
* No waiting period for patients who relapse while receiving standard maintenance therapy
* Patients who relapse on frontline therapy in phases other than maintenance must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Cytotoxic therapy: at least 14 days since the completion of cytotoxic therapy with the exception of hydroxyurea, which is permitted up to 24 hours prior to the start of protocol therapy, or maintenance chemotherapy, or intrathecal chemotherapy (methotrexate strongly preferred) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status
* Biologic (anti-neoplastic) agent: at least 7 days since the completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
* Stem cell transplant or rescue: patient has not had a prior stem cell transplant or rescue
* Patient has not had prior treatment with blinatumomab
* With the exception of intrathecal chemotherapy (methotrexate strongly preferred; cytarabine is permissible) administered at the time of the required diagnostic lumbar puncture to establish baseline CNS status, patient has not received prior relapse-directed therapy (i.e., this protocol is intended as the INITIAL treatment of first relapse)
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: =< 0.6 mg/dL
  * 2 to < 6 years: =< 0.8 mg/dL
  * 6 to < 10 years: =< 1 mg/dL
  * 10 to < 13 years: =< 1.2 mg/dL
  * 13 to < 16 years: =< 1.5 mg/dL (males) and =< 1.4 mg/dL (females)
  * >= 16 years: =< 1.7 mg/dL (males) and =< 1.4 mg/dL (females)
* Direct bilirubin < 3.0 mg/dL
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram
* All patients and/or their parent or legal guardian must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with Philadelphia chromosome positive/breakpoint cluster region protein (BCR)-Abelson murine leukemia viral oncogene homolog 1 (ABL1)+ ALL are not eligible
* Patients with Burkitt leukemia/lymphoma or mature B-cell leukemia are not eligible
* Patients with T-lymphoblastic leukemia (T-ALL)/lymphoblastic lymphoma (T-LL) are not eligible
* Patients with B-lymphoblastic lymphoma (B-LL) are not eligible
* Patients with known optic nerve and/or retinal involvement are not eligible; patients who are presenting with visual disturbances should have an ophthalmologic exam and, if indicated, a magnetic resonance imaging (MRI) to determine optic nerve or retinal involvement
* Patients known to have one of the following concomitant genetic syndromes: Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome
* Patients with known human immunodeficiency virus (HIV) infection
* Patients with known allergy to mitoxantrone, cytarabine, or both etoposide and etoposide phosphate (Etopophos)
* Lactating females who plan to breastfeed
* Patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs; a pregnancy test is required for female patients of childbearing potential
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* Patients with pre-existing significant central nervous system pathology that would preclude treatment with blinatumomab, including: history of severe brain injury, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination/movement disorder, or autoimmune disease with CNS involvement are not eligible; patients with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible; (patients with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved)
* Patients with uncontrolled seizure disorder are not eligible; (patients with seizure disorders that do not require antiepileptic drugs, or are well controlled with stable doses of antiepileptic drugs remain eligible)

Ages: 1 Year to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 669 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2026-09-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Brown, Principal Investigator — Children's Oncology Group
Locations (186):
- United States (166):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (13):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Hogan LE, Bhatla T, Xu X, Gore L, Raetz EA, Bhojwani D, Teachey DT, Hunger SP, Loh ML, Brown PA, Ji L. Severe toxicity and poor efficacy of reinduction chemotherapy are associated with overall poor outcomes in relapsed B-cell acute lymphoblastic leukemia: a report from the Children's Oncology Group AALL1331 trial. Haematologica. 2025 Dec 1;110(12):2930-2941. doi: 10.3324/haematol.2025.287386. Epub 2025 Jun 26. PMID 40568722
- [Derived] Hogan LE, Brown PA, Ji L, Xu X, Devidas M, Bhatla T, Borowitz MJ, Raetz EA, Carroll A, Heerema NA, Zugmaier G, Sharon E, Bernhardt MB, Terezakis SA, Gore L, Whitlock JA, Hunger SP, Loh ML. Children's Oncology Group AALL1331: Phase III Trial of Blinatumomab in Children, Adolescents, and Young Adults With Low-Risk B-Cell ALL in First Relapse. J Clin Oncol. 2023 Sep 1;41(25):4118-4129. doi: 10.1200/JCO.22.02200. Epub 2023 May 31. PMID 37257143
- [Derived] Brown PA, Ji L, Xu X, Devidas M, Hogan LE, Borowitz MJ, Raetz EA, Zugmaier G, Sharon E, Bernhardt MB, Terezakis SA, Gore L, Whitlock JA, Pulsipher MA, Hunger SP, Loh ML. Effect of Postreinduction Therapy Consolidation With Blinatumomab vs Chemotherapy on Disease-Free Survival in Children, Adolescents, and Young Adults With First Relapse of B-Cell Acute Lymphoblastic Leukemia: A Randomized Clinical Trial. JAMA. 2021 Mar 2;325(9):833-842. doi: 10.1001/jama.2021.0669. PMID 33651090
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First relapsed childhood B-Lymphoblastic Leukemia (B-ALL)
Pre-assignment Details: All patients received 4 weeks of Block 1 reinduction chemotherapy. Following reinduction, individuals in the high- and intermediate-risk group were randomized in a 1:1 ratio to receive Arm A or Arm B, and individuals in the low-risk group were randomized in a 1:1 ratio to receive Arm C or Arm D. Patients who fail Arm A had the option to move to Arm: Blinatumomab salvage therapy
Groups:
- Block 1 Induction Therapy: All relapsed B-ALL patients enrolled on AALL1331 for Block 1 induction therapy.
- Arm A (HR and IR Control): Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, and then undergo allogeneic HSCT if eligible. Patients with persistent testicular involvement after Block 1 receive testicular radiation during the Block 2.
- Arm B (HR and IR Blinatumomab); Blinatumomab Salvage Therapy: Patients receive Blinatumomab Block 1 over 5 weeks, Blinatumomab Block 2 over 5 weeks, and then undergo allogeneic HSCT if eligible. Patients with persistent testicular involvement after Block 1 receive testicular radiation during the first block of blinatumomab.
- Arm C (LR Control): Patients receive Block 2 over 4 weeks, Block 3 over 4 weeks, Continuation 1 over 8 weeks, Continuation 2 over 8 weeks, and then Maintenance. CNS3 patients receive chemoradiation post-Maintenance Cycle 1. Patients with persistent testicular involvement after Block 1 receive testicular radiation during Block 2.
- Arm D (LR Blinatumomab): Patients receive Block 2 over 4 weeks, Blinatumomab Cycle 1 over 5 weeks, Continuation 1 over 8 weeks, Blinatumomab Cycle 2 over 5 weeks, Continuation 2 over 8 weeks, Blinatumomab Cycle 3 over 5 weeks, and then Maintenance. CNS3 patients receive chemoradiation post Maintenance Cycle 1. Patients with persistent testicular involvement after Block 1 receive testicular radiation during Block 2.
Period: Block 1 Induction
Arm/Group | Block 1 Induction Therapy | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab) | Arm C (LR Control) | Arm D (LR Blinatumomab) | Blinatumomab Salvage Therapy
Started | 669 | 0 | 0 | 0 | 0 | 0
Completed | 494 | 0 | 0 | 0 | 0 | 0
Not Completed | 175 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 20 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 61 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 65 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Development of significant central nervous system pathology pre-randomization | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Repeat eligibility studies are outside the parameters required for eligibility | 1 | 0 | 0 | 0 | 0 | 0
Period: Post Induction Randomization
Arm/Group | Block 1 Induction Therapy | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab) | Arm C (LR Control) | Arm D (LR Blinatumomab) | Blinatumomab Salvage Therapy
Started | 0 | 109 | 107 | 129 | 127 | 0
Completed | 0 | 14 | 31 | 78 | 79 | 0
Not Completed | 0 | 95 | 76 | 51 | 48 | 0
Not completed — Adverse Event | 0 | 3 | 8 | 4 | 4 | 0
Not completed — Death | 0 | 9 | 2 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 14 | 23 | 18 | 21 | 0
Not completed — Physician Decision | 0 | 43 | 23 | 14 | 14 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 13 | 12 | 7 | 8 | 0
Not completed — Repeat eligibility studies are outside the parameters required for eligibility | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Found to be ineligible for HSCT | 0 | 5 | 8 | 0 | 0 | 0
Not completed — Proceeded to Blinatumomab salvage therapy | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Patient still receiving protocol therapy | 0 | 0 | 0 | 5 | 1 | 0
Period: Blinatumomab Salvage Therapy
Arm/Group | Block 1 Induction Therapy | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab) | Arm C (LR Control) | Arm D (LR Blinatumomab) | Blinatumomab Salvage Therapy
Started | 0 | 0 | 0 | 0 | 0 | 27
Completed | 0 | 0 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 25
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All relapsed B-ALL patients enrolled on AALL1331
Arm/Group | Block 1 Induction Therapy
Number analyzed (Participants) | 669
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 585
  Between 18 and 65 years | 84
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284
  Male | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 221
  Not Hispanic or Latino | 425
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 61
  White | 468
  More than one race | 7
  Unknown or Not Reported | 90
Region of Enrollment [Number; unit: participants]
  Australia | 5
  Canada | 58
  New Zealand | 10
  United States | 596

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) of High-risk (HR) and Intermediate-risk (IR) Relapse Patients
Description: DFS rates of HR and IR relapse B-ALL patients who are randomized following Induction Block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR Randomization). DFS is calculated as the time from randomization to date of first event (treatment failure, relapse, second malignancy, remission death) or date of last contact. Two-year DFS estimates will be calculated from date of randomization for both Arm A and Arm B. Two-sided 95% confidence intervals will be calculated.
Time Frame: Up to 2 years from date of randomization
Population: HR and IR patients randomized per protocol prior to June 30, 2019. This is the cohort of patients who were included in the primary analysis addressing the primary objective on HR/IR patients. Of the total of 216 randomized HR/IR patients, 2 patients with randomization procedure errors and 6 patients randomized after June 30, 2019 were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab)
Number analyzed (Participants) | 103 | 105
percentage of participants | 39.04 [29.13 to 48.81] | 54.44 [44.30 to 63.51]

2. Primary Outcome: Disease Free Survival (DFS) of Low Risk (LR) Relapse Patients
Description: DFS rates of LR relapse B-ALL patients who are randomized following Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization). DFS is calculated as the time from randomization to date of first event (relapse, second malignancy, remission death) or date of last contact. Three-year DFS estimates will be calculated from date of randomization for both Arm C and Arm D. Two-sided 95% confidence intervals will be calculated.
Time Frame: Up to 3 years from date of randomization
Population: LR patients randomized per protocol. This is the cohort of patients who were included in the primary analysis addressing the primary objective on LR patients. Of the total of 256 randomized LR patients, 1 patient was found to be ineligible and was excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C (LR Control) | Arm D (LR Blinatumomab)
Number analyzed (Participants) | 128 | 127
percentage of participants | 58.94 [49.08 to 67.53] | 67.00 [57.36 to 74.94]

3. Secondary Outcome: Overall Survival (OS) of HR and IR Relapse Patients
Description: OS rates of HR and IR relapse B-ALL patients who are randomized following Induction Block 1 chemotherapy to receive either two intensive chemotherapy blocks or two 5-week blocks of blinatumomab (HR/IR Randomization). OS is calculated as the time from randomization to date of death or date of last contact. Two-year OS estimates will be calculated from date of randomization for both Arm A and Arm B. Two-sided 95% confidence intervals will be calculated.
Time Frame: Up to 2 years from date of randomization
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab)
Number analyzed (Participants) | 103 | 105
percentage of participants | 58.40 [47.75 to 67.61] | 71.33 [61.34 to 79.17]

4. Secondary Outcome: Overall Survival (OS) of LR Relapse Patients
Description: OS rates of LR relapse B-ALL patients who are randomized following Block 1 chemotherapy to receive either chemotherapy alone or chemotherapy plus blinatumomab (LR Randomization). OS is calculated as the time from randomization to date of death or date of last contact. Three-year OS estimates will be calculated from date of randomization for both Arm C and Arm D. Two-sided 95% confidence intervals will be calculated.
Time Frame: Up to 3 years from date of randomization
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm C (LR Control) | Arm D (LR Blinatumomab)
Number analyzed (Participants) | 128 | 127
percentage of participants | 88.29 [80.96 to 92.92] | 90.37 [82.63 to 94.77]

5. Other Pre Specified Outcome: Rates of Minimal Residual Disease (MRD) Positivity (> 0.01%)
Description: The rates at the end of Block 2 and Block 3 will be calculated for the randomized arms for HR and IR relapse patients.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Hematologic Complete Remission Rate (for Treatment Failure Patients Not Previously Receiving Blinatumomab)
Description: The observed rate will be calculated among patients with treatment failure who did not previously receive blinatumomab.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: MRD Negativity (< 0.01%) Rate (for Treatment Failure Patients Not Previously Receiving Blinatumomab)
Description: The observed rate will be calculated among patients with treatment failure who did not previously receive blinatumomab.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Proportion of Patients That Proceed to Hematopoietic Stem Cell Transplant (HSCT) After Treatment With Blinatumomab (for Treatment Failure Patients Not Previously Receiving Blinatumomab)
Description: The observed rate will be calculated among patients with treatment failure who did not previously receive blinatumomab.
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Feasibility of Rapid Taper of Immune Suppression for Subset of HSCT Patients With MRD >= 0.01% Pre- and/or Post-HSCT With no Acute Graft Versus Host Disease (aGVHD)
Description: The observed rate of grade III-IV aGVHD among this subset will be calculated with 95% confidence intervals and compared descriptively to target rate.
Time Frame: Up to 10 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Safety of Rapid Taper of Immune Suppression for Subset of HSCT Patients With MRD >= 0.01% Pre- and/or Post-HSCT With no aGVHD Defined as < 5% Rate of Treatment-related Mortality (TRM)
Description: The observed rate of TRM among this subset will be calculated with 95% confidence intervals and compared descriptively to target rate.
Time Frame: Up to 10 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Blinatumomab Pharmacokinetics (PK)
Description: Blinatumomab PK will be evaluated by summarizing blinatumomab steady state concentrations and systemic clearance obtained from non-compartmental analysis. In addition, a population PK approach using a non-linear mixed effect model will also be used to assess blinatumomab PK. Exposure-response analyses will be performed to explore associations among blinatumomab exposure, relevant clinical covariates and clinical measures of safety and efficacy.
Time Frame: Days 2 and 14 of cycle 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years from start of Block 1 to end of protocol therapy
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Groups:
- Blinatumomab Salvarage Therapy: Patients receive Blinatumomab Block 1 over 5 weeks, Blinatumomab Block 2 over 5 weeks, and then undergo allogeneic HSCT if eligible. Patients with persistent testicular involvement after Block 1 receive testicular radiation during the first block of blinatumomab.
Arm/Group | Block 1 Induction Therapy | Arm A (HR and IR Control) | Arm B (HR and IR Blinatumomab) | Arm C (LR Control) | Arm D (LR Blinatumomab) | Blinatumomab Salvarage Therapy
All-Cause Mortality (participants affected / at risk) | 24/661 | 9/109 | 5/107 | 3/129 | 0/127 | 2/27
Serious Adverse Events (participants affected / at risk) | 63/661 | 26/109 | 45/107 | 16/129 | 69/127 | 16/27
Other Adverse Events (participants affected / at risk) | 456/661 | 92/109 | 103/107 | 118/129 | 123/127 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Block 1 Induction Therapy (N=661) | Arm A (HR and IR Control) (N=109) | Arm B (HR and IR Blinatumomab) (N=107) | Arm C (LR Control) (N=129) | Arm D (LR Blinatumomab) (N=127) | Blinatumomab Salvarage Therapy (N=27)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 5 (5) | 3 (3) | 5 (6) | 19 (27) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Death NOS (General disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 10 (10) | 2 (2)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 1 (1)
Sudden death NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 6 (7) | 3 (3)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 11 (12) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 7 (8) | 3 (3) | 2 (2) | 1 (1) | 7 (8) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (2) | 4 (5) | 2 (3) | 5 (5) | 1 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 26 (31) | 10 (11) | 3 (4) | 5 (5) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 5 (5) | 2 (4) | 6 (7) | 4 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 4 (5) | 2 (2) | 5 (6) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 7 (7) | 0 (0)
Stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, specify (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 9 (9) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Block 1 Induction Therapy (N=661) | Arm A (HR and IR Control) (N=109) | Arm B (HR and IR Blinatumomab) (N=107) | Arm C (LR Control) (N=129) | Arm D (LR Blinatumomab) (N=127) | Blinatumomab Salvarage Therapy (N=27)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 70 (134) | 82 (124) | 86 (207) | 95 (236) | 20 (33)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 1 (1) | 4 (6) | 2 (2) | 1 (4)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 191 (204) | 55 (71) | 2 (2) | 78 (165) | 63 (126) | 7 (7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 3 (5) | 1 (1) | 1 (2) | 3 (3) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 4 (6) | 5 (6) | 4 (4) | 6 (6) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 10 (10) | 22 (25) | 28 (37) | 35 (45) | 32 (53) | 9 (9)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 10 (11) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 8 (8) | 4 (5) | 19 (20) | 0 (0) | 0 (0)
Corneal ulcer (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 2 (3) | 3 (4) | 7 (7) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 5 (6) | 4 (5) | 17 (17) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 4 (4) | 4 (4) | 9 (9) | 2 (2) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 18 (18) | 19 (23) | 19 (23) | 30 (35) | 26 (32) | 5 (6)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 5 (5) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 20 (22) | 24 (30) | 23 (28) | 19 (31) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 14 (15) | 20 (27) | 14 (17) | 36 (39) | 23 (26) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (8) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 37 (37) | 52 (63) | 5 (6) | 57 (89) | 42 (48) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (13) | 28 (40) | 34 (46) | 46 (57) | 33 (55) | 11 (14)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2) | 9 (10) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 18 (18) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 7 (8) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 19 (19) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 31 (43) | 23 (29) | 42 (52) | 25 (36) | 9 (11)
Chills (General disorders) | 0 (0) | 7 (9) | 8 (10) | 12 (13) | 12 (12) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 7 (7) | 3 (3) | 3 (3) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 5 (6) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Edema trunk (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 17 (19) | 15 (18) | 29 (39) | 25 (31) | 4 (4)
Fever (General disorders) | 14 (14) | 39 (48) | 56 (76) | 52 (64) | 75 (121) | 17 (34)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 3 (3) | 1 (1) | 7 (14) | 3 (3) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 3 (5) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Localized edema (General disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 3 (4) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 2 (3) | 4 (4) | 6 (7) | 0 (0)
Pain (General disorders) | 11 (13) | 11 (13) | 16 (21) | 18 (28) | 16 (22) | 4 (5)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (6)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 6 (6) | 1 (1) | 9 (11) | 5 (5) | 1 (1)
Anaphylaxis (Immune system disorders) | 5 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 2 (2) | 19 (21) | 0 (0) | 14 (23) | 5 (5)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (3) | 6 (10) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 21 (26) | 8 (11) | 0 (0) | 8 (8) | 5 (7) | 0 (0)
Cecal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 6 (6) | 6 (6) | 0 (0) | 10 (14) | 7 (9) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 115 (150) | 32 (48) | 11 (17) | 56 (97) | 30 (35) | 3 (3)
Infective myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 34 (34) | 10 (12) | 2 (2) | 19 (25) | 12 (26) | 2 (2)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 6 (6) | 1 (1) | 1 (1) | 2 (3) | 1 (2) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (3) | 3 (3) | 2 (3) | 5 (7) | 8 (11) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 5 (5) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 39 (41) | 18 (19) | 0 (0) | 21 (24) | 10 (10) | 0 (0)
Sinusitis (Infections and infestations) | 9 (9) | 3 (3) | 2 (2) | 12 (12) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 12 (12) | 9 (10) | 2 (2) | 13 (15) | 8 (10) | 2 (2)
Small intestine infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 4 (6) | 2 (2) | 0 (0)
Splenic infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (6) | 13 (19) | 5 (5) | 20 (29) | 18 (34) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 10 (11) | 1 (1) | 9 (17) | 8 (10) | 0 (0)
Vulval infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 5 (8) | 3 (4) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomal ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 6 (6) | 10 (11) | 6 (6) | 6 (6) | 3 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 90 (93) | 67 (110) | 76 (107) | 102 (363) | 92 (243) | 17 (23)
Alkaline phosphatase increased (Investigations) | 2 (2) | 18 (25) | 21 (27) | 14 (19) | 15 (22) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 46 (46) | 57 (88) | 58 (78) | 83 (185) | 67 (115) | 15 (21)
Blood bilirubin increased (Investigations) | 44 (46) | 41 (54) | 20 (22) | 61 (117) | 28 (59) | 3 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 5 (7) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 5 (6) | 2 (2) | 13 (15) | 5 (5) | 2 (2)
Ejection fraction decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 11 (11) | 4 (4) | 4 (9) | 1 (1) | 2 (2) | 0 (0)
GGT increased (Investigations) | 13 (13) | 13 (19) | 11 (13) | 14 (21) | 10 (14) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
INR increased (Investigations) | 2 (2) | 6 (8) | 6 (6) | 4 (4) | 1 (1) | 4 (4)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (4) | 7 (15) | 4 (6) | 9 (24) | 2 (2)
Lipase increased (Investigations) | 27 (27) | 5 (5) | 0 (0) | 5 (7) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4) | 37 (64) | 54 (86) | 65 (163) | 72 (181) | 11 (28)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (15) | 62 (103) | 62 (103) | 87 (232) | 90 (218) | 19 (30)
Platelet count decreased (Investigations) | 10 (10) | 71 (122) | 49 (68) | 81 (185) | 71 (125) | 21 (35)
Serum amylase increased (Investigations) | 7 (7) | 6 (6) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Weight gain (Investigations) | 1 (1) | 3 (3) | 5 (6) | 6 (11) | 9 (21) | 2 (2)
Weight loss (Investigations) | 10 (10) | 8 (9) | 5 (6) | 12 (14) | 9 (9) | 2 (2)
White blood cell decreased (Investigations) | 7 (7) | 64 (116) | 75 (128) | 81 (252) | 92 (244) | 17 (28)
Acidosis (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 41 (41) | 21 (26) | 14 (17) | 30 (41) | 17 (22) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 12 (12) | 8 (8) | 3 (3) | 11 (13) | 9 (9) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 8 (10) | 4 (4) | 5 (6) | 4 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 109 (110) | 37 (54) | 47 (71) | 51 (74) | 53 (118) | 15 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 11 (11) | 12 (14) | 10 (11) | 15 (16) | 10 (10) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (2) | 10 (11) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 19 (22) | 9 (10) | 17 (22) | 7 (12) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 19 (19) | 12 (13) | 3 (3) | 7 (7) | 8 (12) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 41 (42) | 52 (79) | 55 (70) | 58 (82) | 49 (83) | 14 (21)
Hypocalcemia (Metabolism and nutrition disorders) | 32 (33) | 47 (68) | 33 (42) | 48 (64) | 44 (66) | 11 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 19 (22) | 9 (9) | 12 (14) | 3 (5) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 76 (76) | 54 (79) | 39 (50) | 61 (112) | 55 (93) | 13 (17)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 29 (37) | 18 (22) | 31 (36) | 15 (20) | 11 (11)
Hyponatremia (Metabolism and nutrition disorders) | 57 (59) | 31 (38) | 29 (39) | 35 (44) | 23 (34) | 8 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 50 (50) | 24 (31) | 24 (28) | 32 (35) | 15 (21) | 9 (13)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (2) | 3 (4) | 2 (3) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 6 (7) | 3 (4) | 4 (5) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (12) | 15 (19) | 16 (21) | 25 (28) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6) | 3 (4) | 6 (6) | 4 (4) | 4 (4)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (3) | 6 (6) | 5 (5) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 4 (5) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 8 (9) | 9 (10) | 8 (11) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 3 (3) | 4 (4) | 7 (7) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 17 (22) | 15 (21) | 15 (18) | 26 (37) | 8 (10)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 7 (8) | 8 (8) | 5 (6) | 11 (11) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 11 (12) | 20 (26) | 36 (54) | 36 (53) | 56 (90) | 11 (14)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (3)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 6 (6) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 9 (11) | 4 (4) | 8 (11) | 4 (6) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7) | 9 (10) | 8 (9) | 3 (4) | 7 (8) | 4 (4)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 9 (11) | 4 (4) | 22 (32) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 2 (2) | 6 (7) | 2 (5) | 6 (8) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (5) | 11 (13) | 11 (12) | 14 (21) | 4 (4)
Confusion (Psychiatric disorders) | 2 (2) | 3 (3) | 7 (7) | 0 (0) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 4 (5) | 7 (10) | 7 (12) | 5 (9) | 1 (1)
Euphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (5) | 3 (3) | 8 (12) | 7 (8) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 5 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 7 (7) | 1 (1) | 4 (4) | 4 (4) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (6) | 5 (7) | 6 (10) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3) | 4 (4) | 1 (2) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 18 (24) | 12 (16) | 27 (32) | 30 (37) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 3 (3) | 9 (10) | 6 (6) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (8) | 1 (1) | 18 (19) | 5 (5) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (13) | 1 (1) | 21 (21) | 9 (9) | 2 (3)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 3 (5) | 14 (15) | 16 (19) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 1 (1) | 6 (7) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 3 (3) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 3 (10) | 2 (3) | 5 (8) | 2 (4)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 4 (5) | 10 (11) | 12 (13) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (7) | 9 (12) | 6 (7) | 13 (19) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 6 (7) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7) | 7 (9) | 5 (5) | 15 (18) | 2 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (8) | 11 (12) | 20 (26) | 16 (17) | 22 (26) | 3 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7) | 10 (13) | 11 (11) | 9 (11) | 3 (3)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (4) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 14 (17) | 2 (2)
Hematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 22 (23) | 24 (33) | 18 (26) | 27 (34) | 15 (23) | 10 (12)
Hypotension (Vascular disorders) | 30 (30) | 16 (17) | 18 (25) | 21 (32) | 33 (49) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02101853/Prot_SAP_000.pdf